CLINICAL TRIAL: NCT00549172
Title: Efficacy of Arthroscopic Partial Resection for the Degenerative Tear of the Medial Meniscus of a Knee
Brief Title: Arthroscopy in the Treatment of Degenerative Medial Meniscus Tear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University (Other)
Collaborators: Helsinki University Central Hospital (Other); Kuopio University Hospital (Other); Turku University Hospital (Other Government); Central Finland Hospital District (Other)
Responsible Party: Principal Investigator, Raine Sihvonen, Principal Investigator, Tampere University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R06157
Record Dates: First submitted 2007-10-24; First posted 2007-10-25 (Estimated); Results first posted 2015-03-23 (Estimated); Last update posted 2023-01-13 (Actual); Status verified 2022-12

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis, Knee; Arthroscopic Surgery; Menisci, Medial; Placebo Effect; Treatment Efficacy
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Operative (O) (Active Comparator): Partial resection of degenerative tear of medial meniscus
  Interventions: Procedure: Operative (partial arthroscopy)
- Conservative (K) (Sham Comparator): Arthroscopy (diagnostic)
  Interventions: Procedure: Conservative (diagnostic arthroscopy)

INTERVENTIONS:
Procedure: Operative (partial arthroscopy) — Partial arthroscopic resection of degenerative rupture of the medial meniscus
  Arms: Operative (O)
Procedure: Conservative (diagnostic arthroscopy) — Diagnostic arthroscopy
  Arms: Conservative (K)

SUMMARY:
Degenerative meniscal tears are the most common etiology for knee pain, swelling and loss of function. Partial arthroscopic meniscectomy is the most common orthopaedic procedure to treat meniscal tears. Improvements have been reported both after arthroscopy and with conservative treatment, however no direct comparison exist. Accordingly, the aim of this study is to assess the efficacy of arthroscopic partial meniscectomy for the treatment of degenerative tear of medial meniscus of the knee using a double-blind, placebo controlled, randomised trial.

DETAILED DESCRIPTION:
Middle-aged men and women with degenerative meniscal tears constitute a large group of patients presenting with knee pain, sometimes accompanied with swelling and loss of function. Many meniscal tears occur without a trauma in physically active individuals as well as in older people and could be a part of early osteoarthritis. Partial arthroscopic meniscectomy is the most common orthopaedic procedure and is used to treat patients with meniscal tears. Many patients report improvement after arthroscopy referring especially to reduced knee pain, better knee function and improved quality of life. However, similar results have also been obtained with conservative treatment (physical therapy) of patients with degenerative meniscal tears. Accordingly, the aim of this study is to assess the efficacy of arthroscopic partial meniscectomy for the treatment of degenerative tear of medial meniscus of the knee using a double-blind, placebo controlled, randomised trial. The outcome of arthroscopic partial meniscectomy (vs. sham surgery) is assessed using the Lysholm knee score and pain at rest and activity (VAS) at 2, 6 and 12 months after the operation. In addition, the functional outcome is assessed using the WOMET knee score (a disease-specific quality of life -knee score development on the assessment of meniscal pathology), the general quality of life score (15-D), and cost-effectiveness analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 35 to 65 years of age.
2. A pain located on the medial joint line of the knee that has persistent at least for 3 months.
3. Pain that can be provoked by palpation or compression of the joint line or a positive McMurray sign.
4. Tear of the medial meniscus on MRI.
5. Degenerative rupture of the medial meniscus confirmed at arthroscopy.

Exclusion Criteria:

1. Acute, trauma-induced onset of symptoms.
2. Locking or painful snapping of the knee joint.
3. A surgical operation performed on the affected knee.
4. Osteoarthritis of the medial compartment of the knee (determined by clinical criteria of the ACR).
5. Osteoarthritis on knee radiographs (Kellgren-Lawrence > 1).
6. Acute (within the previous year) fractures of the knee.
7. Decreased range of motion of the knee.
8. Instability of the knee.
9. MRI assessment showing a tumor or any other complaint requiring surgical or other means of treatment.
10. Arthroscopic assessment showing anything other than a degenerative tear of the medial meniscus requiring surgical intervention.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2007-10; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teppo LN Jarvinen, MD, PhD, Study Chair — Tampere University; Raine TA Sihvonen, MD, Principal Investigator — Tampere City Hospital; Mika Paavola, MD, PhD, Study Director — University of Helsinki; Antti Malmivaara, MD, PhD, Study Director — University of Helsinki
Locations (5):
- Finland (5):
  - Helsinki Central Hospital, Helsinki
  - Central Finland Hospital District, Jyväskylä
  - Kuopio University Hospital, Kuopio
  - Hatanpää City Hospital, Tampere
  - Turku University Hospital, Turku

REFERENCES:
- [Derived] Sillanpaa N, Iivanainen M, Turkiewicz A, Sihvonen R, Paavola M, Taimela S, Jarvinen TLN, Englund M. Effect of arthroscopic partial meniscectomy on structural degeneration of the knee - A 5-year MRI-based follow-up of the placebo-surgery controlled FIDELITY (Finnish Degenerative Meniscus Lesion Study) trial. Osteoarthritis Cartilage. 2025 Feb;33(2):276-282. doi: 10.1016/j.joca.2024.09.003. Epub 2024 Sep 12. PMID 39277028
- [Derived] Kalske R, Kiadaliri A, Sihvonen R, Englund M, Turkiewicz A, Paavola M, Malmivaara A, Itala A, Joukainen A, Nurmi H, Toivonen P, Taimela S, Jarvinen TLN; FIDELITY (Finnish Degenerative Meniscal Lesion Study) Investigators. Arthroscopic Partial Meniscectomy for a Degenerative Meniscus Tear Is Not Cost Effective Compared With Placebo Surgery: An Economic Evaluation Based on the FIDELITY Trial Data. Clin Orthop Relat Res. 2024 Sep 1;482(9):1523-1533. doi: 10.1097/CORR.0000000000003094. Epub 2024 May 7. PMID 38905520
- [Derived] Sihvonen R, Paavola M, Malmivaara A, Itala A, Joukainen A, Kalske J, Nurmi H, Kumm J, Sillanpaa N, Kiekara T, Turkiewicz A, Toivonen P, Englund M, Taimela S, Jarvinen TLN; FIDELITY (Finnish Degenerative Meniscus Lesion Study) Investigators. Arthroscopic partial meniscectomy for a degenerative meniscus tear: a 5 year follow-up of the placebo-surgery controlled FIDELITY (Finnish Degenerative Meniscus Lesion Study) trial. Br J Sports Med. 2020 Nov;54(22):1332-1339. doi: 10.1136/bjsports-2020-102813. Epub 2020 Aug 27. PMID 32855201
- [Derived] Sihvonen R, Kalske R, Englund M, Turkiewicz A, Toivonen P, Taimela S, Jarvinen TLN; Finnish Degenerative Meniscal Lesion Study (FIDELITY) Investigators. Statistical analysis plan for the 5-year and 10-year follow-up assessments of the FIDELITY trial. Trials. 2020 Jan 14;21(1):76. doi: 10.1186/s13063-019-3833-2. PMID 31937344
- [Derived] Sihvonen R, Englund M, Turkiewicz A, Jarvinen TL; Finnish Degenerative Meniscal Lesion Study Group. Mechanical Symptoms and Arthroscopic Partial Meniscectomy in Patients With Degenerative Meniscus Tear: A Secondary Analysis of a Randomized Trial. Ann Intern Med. 2016 Apr 5;164(7):449-55. doi: 10.7326/M15-0899. Epub 2016 Feb 9. PMID 26856620
- [Derived] Sihvonen R, Paavola M, Malmivaara A, Itala A, Joukainen A, Nurmi H, Kalske J, Jarvinen TL; Finnish Degenerative Meniscal Lesion Study (FIDELITY) Group. Arthroscopic partial meniscectomy versus sham surgery for a degenerative meniscal tear. N Engl J Med. 2013 Dec 26;369(26):2515-24. doi: 10.1056/NEJMoa1305189. PMID 24369076
- [Derived] Sihvonen R, Paavola M, Malmivaara A, Jarvinen TL. Finnish Degenerative Meniscal Lesion Study (FIDELITY): a protocol for a randomised, placebo surgery controlled trial on the efficacy of arthroscopic partial meniscectomy for patients with degenerative meniscus injury with a novel 'RCT within-a-cohort' study design. BMJ Open. 2013 Mar 9;3(3):e002510. doi: 10.1136/bmjopen-2012-002510. PMID 23474796

RESULTS

PARTICIPANT FLOW:
Groups:
- Operative (O): Partial resection of degenerative tear of medial meniscus
  Operative (partial arthroscopy): Partial arthroscopic resection of degenerative rupture of the medial meniscus
  n=70
- Conservative (K): Arthroscopy (diagnostic)
  Conservative (diagnostic arthroscopy): Diagnostic arthroscopy
  n=76
Period: Overall Study
Arm/Group | Operative (O) | Conservative (K)
Started | 70 | 76
Completed | 70 | 76
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Age, Sex, Weight, Height, BMI, Duration of medial knee pain, Type of onset of symptoms, Radiographic assessment (Kellfren-Lawrence), Clinical meniscal tests
Groups:
- Total: Total of all reporting groups
Arm/Group | Operative (O) | Conservative (K) | Total
Number analyzed (Participants) | 70 | 76 | 146
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (7) | 52 (7) | 52 (7)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 70 | 76 | 146
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 29 | 57
  Male | 42 | 47 | 89
Region of Enrollment [Number; unit: participants]
  Finland | 70 | 76 | 146

OUTCOME MEASURES:

1. Primary Outcome: The Lysholm Knee Score
Description: The Lysholm knee score is based on an eight-item questionnaire designed to evaluate knee function and symptoms in activities of daily living. Scores range from 0 to 100; higher scores indicate less severe symptoms.
Time Frame: One year
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Operative (O) | Conservative (K)
Number analyzed (Participants) | 70 | 76
units on a scale | 82.2 [78.4 to 85.9] | 83.4 [80.3 to 86.5]

2. Primary Outcome: Pain After Exercise (VAS)
Description: Knee pain after exercise (during the preceding week) was assessed on a rating scale of 0 to 10, with 0 denoting no pain and 10 denoting extreme pain.
Time Frame: One year
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Operative (O) | Conservative (K)
Number analyzed (Participants) | 70 | 76
units on a scale | 2.7 [2.1 to 3.3] | 2.9 [2.3 to 3.4]

3. Primary Outcome: WOMET (Western Ontario Meniscal Tear -Disease Specific Quality of Life -Assessment Tool)
Description: The Western Ontario Meniscal Evaluation Tool (WOMET) contains 16 items addressing three domains: 9 items addressing physical symptoms; 4 items addressing disabilities with regard to sports, recreation, work, and lifestyle; and 3 items addressing emotions. The score indicates the percentage of a normal score; therefore, 100 is the best possible score, and 0 is the worst possible score.
Time Frame: One year
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Operative (O) | Conservative (K)
Number analyzed (Participants) | 70 | 76
units on a scale | 81.0 [76.1 to 85.9] | 79.9 [75.1 to 84.7]

4. Secondary Outcome: 15-D (General Quality of Life -Assessment Tool)
Description: The 15D instrument is a generic health-related quality-of-life instrument comprising 15 dimensions. The maximum 15D score is 1 (full health), and the minimum score is 0 (death).
Time Frame: One year
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Operative (O) | Conservative (K)
Number analyzed (Participants) | 70 | 76
units on a scale | 0.94 [0.92 to 0.95] | 0.92 [0.90 to 0.93]

5. Secondary Outcome: Pain at Rest (VAS)
Description: Knee pain at rest (during the preceding week) was assessed on a rating scale of 0 to 10, with 0 denoting no pain and 10 denoting extreme pain.
Time Frame: One year
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Operative (O) | Conservative (K)
Number analyzed (Participants) | 70 | 76
units on a scale | 1.6 [1.0 to 2.1] | 1.9 [1.4 to 2.5]

6. Secondary Outcome: Cost Effectiveness
Description: Cost effectiveness data comparing arthroscopic partial meniscectomy and diagnostic arthroscopy. Costs are based on healthcare utilisation and sickness absence.
Time Frame: 1 and 2 years
Reporting Status: Not Posted, anticipated posting 2023-11

ADVERSE EVENTS:
Arm/Group | Operative (O) | Conservative (K)
Serious Adverse Events (participants affected / at risk) | 1/70 | 0/76
Other Adverse Events (participants affected / at risk) | 0/70 | 0/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Operative (O) (N=70) | Conservative (K) (N=76)
Serious adverse event (Infections and infestations) | 1 (1) | 0 (0) — A deep infection of the index knee 4 months after surgery

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No